CLINICAL TRIAL: NCT05150561
Title: The Prevalence and the Prognostic Value of Sarcopenia Among Patients With Haematological Cancer Diseases - A Prospective Observational Cohort Study.
Brief Title: Muscle Dysfunction in Patients With Haematological Diseases
Status: Active, not recruiting | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Jan Christensen, Senior Researcher, Rigshospitalet, Denmark
Other Study IDs: MuscleLab2020
Record Dates: First submitted 2021-11-08; First posted 2021-12-09 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Hematologic Diseases; Acute Myeloid Leukemia; Acute Lymphoid Leukemia; Myelodysplastic Syndromes; Lymphoma
Keywords: Hematological cancer diseases; Muscle mass; Muscle strength; Complications; Patient reported outcomes; Physical function
MeSH Terms: conditions — Hematologic Diseases; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Myelodysplastic Syndromes; Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Cohort I - Patients newly diagnosed with malignant lymphoma (n=72): These patients will undergo two assessments: A baseline-assessment prior to treatment for the hematologic cancer disease and a follow-up assessment at 6 months after treatment start
- Cohort II - Patients newly diagnosed with acute leukaemia (n=72): These patients will undergo two assessments: A baseline-assessment prior to treatment for the hematologic cancer disease and a follow-up assessment at 6 months after treatment start
- Cohort III - Patients newly diagnosed with multiple myeloma (n=72): These patients will undergo two assessments: A baseline-assessment prior to treatment for the hematologic cancer disease and a follow-up assessment at 6 months after treatment start

SUMMARY:
PURPOSE: To evaluate the prevalence and prognostic value of sarcopenia in patients diagnosed with hematological cancer diseases.

DETAILED DESCRIPTION:
Some patients diagnosed with malignant hematological diseases are faced with poor prognosis and thus must undergo a demanding course of treatment associated with severe deconditioning potentially leading to worse prognostic outcomes. It is currently not well-described, to what extend patients body composition at the point of diagnoses should be part of standard clinical evaluation in order to optimize therapy-efficacy. Recent findings suggest that pathophysiological alterations in skeletal muscle mass and function can have significant implications for the risk of disease progression and long-term prognosis.

ELIGIBILITY:
Inclusion Criteria:

• Patients diagnosed with malignant lymphomas, acute leukaemia and multiple myeloma referred to treatment at the Department of Haematology, Rigshospitalet.

Exclusion Criteria:

* Age: <18
* Pregnancy
* Physical or mental disabilities precluding test of muscle function
* Inability to read and understand Danish.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with malignant lymphomas, acute leukaemia and multiple myeloma referred to treatment.
Sampling Method: Non-Probability Sample
Enrollment: 216 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Change in Whole body Lean body Mass | Baseline and 6 months after treatment start
  Dual-energy X-ray Absorptiometry (DXA) scan

SECONDARY OUTCOMES:
Hospitalization duration | 1 year post treatment
  Total number days in hospital
Disease free survival | 1 year post treatment
  Risk of disease progression
Overall survival | 1 year post treatment
  Risk of mortality from any-cause
Change in appendicular lean mass | Baseline and 6 after treatment start
  Dual-energy X-ray Absorptiometry (DXA) scan
Change in whole body fat percentage | Baseline and 6 months after treatment start
  Dual-energy X-ray Absorptiometry (DXA) scan
Change in visceral fat mass | Baseline and 6 months after treatment start
  Dual-energy X-ray Absorptiometry (DXA) scan
Change in bone mineral density | Baseline and 6 months after treatment start
  Dual-energy X-ray Absorptiometry (DXA) scan
Change in bone mineral content | Baseline and 6 months after treatment start
  Dual-energy X-ray Absorptiometry (DXA) scan
Change in walking capacity | Baseline and 6 months after treatment start
  Maximum 10 meter walking speed
Change in lower body physical function | Baseline and 6 months after treatment start
  30 seconds Sit-To-Stand test
Change in maximum leg power | Baseline and 6 months after treatment start
  Leg extensor power test (Nottingham Power Rig)
Change in hand grip strength | Baseline and 6 months after treatment start
  Maximum strength test by handgrip dynamometer
Change in inflammation markers | Baseline and 6 months after treatment start
  Blood values are registered from the patients hospital record in relation to assessments. C-reactive protein (CRP) and leucocytes are registered as they are inflammation markers.
Change in creatinine | Baseline and 6 months after treatment start
  Blood values are registered from the patients hospital record in relation to assessments. Creatinine is registered due to their relation to muscle strength..
Change in hemoglobin | Baseline and 6 months after treatment start
  Blood values are registered from the patients hospital record in relation to assessments. Hemoglobin is registered due to their relation to muscle strength.
Change in body fat percentage | Baseline and 6 months after treatment start
  Bioelectrical Impedance Analyzer
Change in fat mass | Baseline and 6 months after treatment start
  Bioelectrical Impedance Analyzer
Change in fat-free mass | Baseline and 6 months after treatment start
  Bioelectrical Impedance Analyzer
Change in muscle mass | Baseline and 6 months after treatment start
  Bioelectrical Impedance Analyzer
Change in bone mass | Baseline and 6 months after treatment start
  Bioelectrical Impedance Analyzer
Change in total body water | Baseline and 6 months after treatment start
  Bioelectrical Impedance Analyzer
Change in health-related quality of life | Baseline and 6 months after treatment start
  European Organisation for Research and Treatment of Cancer Quality of LifeQuestionnaire, Version 3.0 Scores range from 0 to 100; a higher score represents a higher ("better") level of functioning, or a higher ("worse") level of symptoms.
Change in physical activity level | Baseline and 6 months after treatment start
  The International Physical Activity Questionnaires, short form. The Questionnaires covers the frequency and duration of vigorous, moderate, and walking activities over the last 7 days, as well as a single-item question on weekday sitting. Using the instrument's scoring protocol, total weekly physical activity can be calculated to three levels of physical activity and the interpretation of the questionnaire can be categorized in low, moderate and high physical activity, based on the stated time and Metabolic Equivalent of Task (METs min/week) used in different types of activities.

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No
Not provided